CLINICAL TRIAL: NCT00810849
Title: A Trial of Adjunctive Prednisolone and Mycobacterium w Immunotherapy in Tuberculous Pericarditis
Acronym: IMPI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Principal Investigator, Bongani M Mayosi, Professor of Medicine, University of Cape Town
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMPI-TRIAL1
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Tuberculous Pericarditis
Keywords: Tuberculosis, pericardium
MeSH Terms: conditions — Pericarditis, Tuberculous | interventions — Prednisolone; Methylprednisolone; Immuvac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisolone (Placebo Comparator): Six-week tapering course of prednisolone and those assigned to the prednisolone control arm will receive the same number of identically-coated placebo tablets.
  Interventions: Drug: Prednisolone
- Mycobacterium w (Placebo Comparator): Patients enrolled in the Mycobacterium w experimental arm will receive 5 doses of 0.1 ml of the vaccine intradermally (on enrolment, at 2 weeks, 4 weeks, 6 weeks, and 3 months).
  Interventions: Biological: Mycobacterium w immunotherapy

INTERVENTIONS:
Drug: Prednisolone — Prednisolone and placebo will be supplied as 5 mg identical tablets and given at a dosage of 120 mg/day in the first week, followed by 90 mg/day in the second week, 60 mg/day in the third week, 30 mg/day in the fourth week, 15 mg/day in the fifth week, and 5 mg/day in the sixth week.
  Other Names: Medrol tablets
  Arms: Prednisolone
Biological: Mycobacterium w immunotherapy — Patients enrolled in the Mycobacterium w experimental arm will receive 5 doses of 0.1 ml of the vaccine intradermally (on enrolment, at 2 weeks, 4 weeks, 6 weeks, and 3 months). Patients in the control arm of the Mycobacterium w comparison will receive a similar regime of placebo injections of normal saline in identically-packaged vials.
  Other Names: Immuvac
  Arms: Mycobacterium w

SUMMARY:
Human immunodeficiency virus (HIV) infection puts people at risk of opportunistic infections, such as tuberculosis. In Africa, the HIV epidemic has resulted in an increase in the number of cases of tuberculosis affecting various parts of the body, including the membrane surrounding the heart (i.e., pericardium). Pericardial tuberculosis is a serious form of tuberculosis that results in the death or disability of 1 in 2 affected people despite the use of antituberculosis medication. It has been suggested that the addition of corticosteroids to the antituberculosis medication could result in the reduction of the number of deaths caused by the disease, but this proposal remains to be confirmed in appropriately designed clinical trials. Similarly, vaccination with the Mycobacterium w injection is also proposed as a possible way of reducing the damage caused by the tuberculosis infection of the heart. The investigators are proposing to conduct a clinical trial in which people who are on antituberculosis treatment for pericardial tuberculosis will be randomly allocated to receive either prednisolone or a matching placebo tablet, or Mycobacterium w injection or placebo injection. The number of people who die or who develop hardening of the pericardium with compression of the heart (called pericardial constriction) or who need emergency evacuation of the pericardial fluid from pericardial sac for severe compression (called tamponade) will be compared in each group to determine whether the use of corticosteroids or Mycobacterium w injection is safe and results in reduction in the death rate. If corticosteroids and Mycobacterium w are shown to safely reduce the death rate, then they will be recommended for use in all patients with tuberculosis of the pericardium in the future.

DETAILED DESCRIPTION:
Summary of research proposal Tuberculous pericarditis is one of the most severe forms of infection with Mycobacterium tuberculosis, causing death or cardiac disability in nearly half of those affected in spite of antituberculosis chemotherapy. Attenuation of the inflammatory response in tuberculous pericarditis may improve outcome by reducing the likelihood of cardiac tamponade and pericardial constriction. A meta-analysis of all randomized controlled trials of corticosteroids for tuberculous pericarditis showed a trend towards reduction of mortality, but the studies were too small to confirm any effect on survival. Concern remains that corticosteroids might increase the frequency of opportunistic infections and cancers in patients infected with the Human Immunodeficiency Virus (HIV). In addition to the promising but inconclusive evidence on adjunctive steroids, there is preliminary evidence suggesting that repeated doses of Mycobacterium w immunotherapy may reduce the inflammation associated with extrapulmonary tuberculosis and increase the CD4 cell count in people infected with HIV. These early observations remain to be tested in a large randomized trial with the hard endpoint of mortality.

The Investigation of the Management of Pericarditis in Africa (IMPI [pronounced as 'ee-mp-ee', for Zulu warriors]) Trial will assess effectiveness and safety of oral prednisolone or placebo and Mycobacterium w immunotherapy or placebo in 1400 patients with tuberculous pericardial effusion. This trial will also determine the feasibility of conducting a large-scale multicentre clinical trial in patients with tuberculous pericarditis in sub-Saharan Africa.

Hypothesis: We hypothesize that patients with suspected tuberculous pericarditis randomized to adjunctive oral prednisolone for 6 weeks will have a 30% reduction in mortality compared to placebo, and that patients randomized to Mycobacterium w injections for 6 months will have a better survival compared to placebo.

Objectives: The primary objectives of the IMPI Trial are: a) to determine the effectiveness of oral prednisolone and Mycobacterium w immunotherapy in reducing the composite outcome of death, constriction or pericardial drainage for cardiac tamponade in patients with tuberculous pericardial effusion, b) to assess the safety and interactive effects of the co-administration of prednisolone and Mycobacterium w immunotherapy, and c) to demonstrate the feasibility of conducting a study in patients with tuberculous pericardial effusion in sub-Saharan Africa, and establish the infrastructure for conducting the full-scale IMPI trial in an internal pilot phase of the first 200 participants.

If the internal pilot phase is positive, all the patients will be rolled-over into the full-scale IMPI trial. The first occurrence of death will be recorded to improve estimates of outcomes for the full-scale trial. Secondary outcomes of the full-scale trial will include: 1) constriction, 2) rate of occurrence of cardiac tamponade requiring pericardiocentesis, 3) rate of resolution of pericardial effusion, 4) improvement in functional class.

Study Design: IMPI is a randomized double-blind placebo-controlled 2x2 factorial pilot trial that will enroll 1400 patients from multiple centres in Kenya, Malawi, Mozambique, Nigeria, Sierra Leone, South Africa, Uganda and Zimbabwe. Patients with tuberculous pericarditis who fulfill the inclusion criteria will be randomly assigned to receive oral prednisolone or placebo for 6 weeks and Mycobacterium w injection or placebo for 6 months. Patients will be followed closely during the intervention period (at weeks 2, 4, 6, and months 3 and 6). Six-monthly follow-up will be performed thereafter for up to two years. The recruitment of the 1400 patients will be performed over 54 months, with a minimum follow-up period of 6 months for the last participants recruited in the trial. The Population Health Research Institute at McMaster University will manage and coordinate the study in association with the IMPI Project Office that is located in the Department of Medicine, Groote Schuur Hospital, Cape Town, South Africa.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted with suspected tuberculous pericarditis will be eligible if they meet all three of the following criteria:

1. A confirmed pericardial effusion on echocardiography;
2. Evidence of definite or probable tuberculous pericarditis; and
3. Within 1 week of starting of antituberculosis treatment.

Exclusion Criteria:

1. Presence of an alternative cause of pericardial disease, e.g., penetrating chest trauma in the previous 12 months and malignancy.
2. Use of corticosteroids within the previous month.
3. Hypersensitivity or allergy to the Mycobacterium w vaccine.
4. Pregnancy.
5. Age < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2008-12; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Composite end-point of death, constriction, or cardiac tamponade requiring pericardial drainage. | Two years

SECONDARY OUTCOMES:
Safety of immunomodulatory treatment | Two years
The secondary efficacy outcomes are the individual components of the composite primary outcome (i.e., death, constriction, and cardiac tamponade requiring pericardiocentesis), and all-cause hospitalization. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Salim Yusuf, M.D., Study Chair — Population Health Research Institute, McMaster University, Hamilton, Canada
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Cape, South Africa

REFERENCES:
- [Background] Mayosi BM, Ntsekhe M, Bosch J, Pogue J, Gumedze F, Badri M, Jung H, Pandie S, Smieja M, Thabane L, Francis V, Thomas KM, Thomas B, Awotedu AA, Magula NP, Naidoo DP, Damasceno A, Banda AC, Mutyaba A, Brown B, Ntuli P, Mntla P, Ntyintyane L, Ramjee R, Manga P, Kirenga B, Mondo C, Russell JB, Tsitsi JM, Peters F, Essop MR, Barasa AF, Mijinyawa MS, Sani MU, Olunuga T, Ogah O, Adebiyi A, Aje A, Ansa V, Ojji D, Danbauchi S, Hakim J, Matenga J, Yusuf S. Rationale and design of the Investigation of the Management of Pericarditis (IMPI) trial: a 2 x 2 factorial randomized double-blind multicenter trial of adjunctive prednisolone and Mycobacterium w immunotherapy in tuberculous pericarditis. Am Heart J. 2013 Feb;165(2):109-15.e3. doi: 10.1016/j.ahj.2012.08.006. Epub 2012 Dec 13. PMID 23351812
- [Derived] Mayosi BM, Ntsekhe M, Bosch J, Pandie S, Jung H, Gumedze F, Pogue J, Thabane L, Smieja M, Francis V, Joldersma L, Thomas KM, Thomas B, Awotedu AA, Magula NP, Naidoo DP, Damasceno A, Chitsa Banda A, Brown B, Manga P, Kirenga B, Mondo C, Mntla P, Tsitsi JM, Peters F, Essop MR, Russell JB, Hakim J, Matenga J, Barasa AF, Sani MU, Olunuga T, Ogah O, Ansa V, Aje A, Danbauchi S, Ojji D, Yusuf S; IMPI Trial Investigators. Prednisolone and Mycobacterium indicus pranii in tuberculous pericarditis. N Engl J Med. 2014 Sep 18;371(12):1121-30. doi: 10.1056/NEJMoa1407380. Epub 2014 Sep 1. PMID 25178809